CLINICAL TRIAL: NCT03699644
Title: Multimodal Ocular Imaging in Neurodegeneration
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Cagri Besirli, Associate Professor of Ophthalmology, University of Michigan
Other Study IDs: HUM00146956
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Disease; Alzheimer Dementia; Frontotemporal Dementia
Keywords: FTD; Dementia; Retina
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Dementia | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography; Fluorescein Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Control: Healthy controls will undergo a single magnetic resonance imaging (MRI) and PET (positron emission tomography) scan of the brain. In addition, all healthy controls will receive a comprehensive ophthalmic examination as well as undergo photography and imaging of the eye.
  Interventions: Device: Spectral-Domain Optical Coherence Tomography (SD-OCT); Device: Magnetic Resonance Imaging (MRI); Device: Positron Emission Tomography (PET); Diagnostic Test: Comprehensive Ophthalmic Examination; Device: Fundus Photography
- Alzheimer's Dementia: Subjects with Alzheimer's Dementia will undergo a single magnetic resonance imaging (MRI) and PET (positron emission tomography) scan of the brain. In addition, all subjects with Alzheimer's Dementia will receive a comprehensive ophthalmic examination as well as undergo photography and imaging of the eye.
  Interventions: Device: Spectral-Domain Optical Coherence Tomography (SD-OCT); Device: Magnetic Resonance Imaging (MRI); Device: Positron Emission Tomography (PET); Diagnostic Test: Comprehensive Ophthalmic Examination; Device: Fundus Photography
- Frontotemporal Dementia: Subjects with Frontotemporal Dementia will undergo a single magnetic resonance imaging (MRI) and PET (positron emission tomography) scan of the brain. In addition, subjects with Frontotemporal Dementia will receive a comprehensive ophthalmic examination as well as undergo photography and imaging of the eye.
  Interventions: Device: Spectral-Domain Optical Coherence Tomography (SD-OCT); Device: Magnetic Resonance Imaging (MRI); Device: Positron Emission Tomography (PET); Diagnostic Test: Comprehensive Ophthalmic Examination; Device: Fundus Photography

INTERVENTIONS:
Device: Spectral-Domain Optical Coherence Tomography (SD-OCT) — Each participant in this study will undergo Optical coherence tomography (OCT), a non-invasive imaging test of the eye, one time. OCT uses light waves to take cross-section pictures of the retina, which are generated using scattered light waves.
  Other Names: Imaging of the Eye
Device: Magnetic Resonance Imaging (MRI) — Each participant in this study will undergo a single Magnetic resonance imaging (MRI) scan, a scanning technique for creating detailed images of the human body. The scan uses a magnetic field and radio waves to generate images of the brain.
Device: Positron Emission Tomography (PET) — Each participant in this study will undergo a single Positron emission tomography (PET) scan of the brain. PET is a nuclear medicine functional imaging technique that is used to observe metabolic processes in the brain as an aid to the diagnosis of disease using the combination of a radioactive tracer, camera, and a computer.
Diagnostic Test: Comprehensive Ophthalmic Examination — Each participant in this study will receive one comprehensive eye examination which will be performed by a licensed ophthalmologist at the University of Michigan. This examination will include the assessment of the participant's visual acuity, a slit lamp examination which will look at the anterior and posterior tissues of the eye including the retina using various lights and lenses, and intraocular pressures.
  Other Names: Comprehensive Eye Examination
Device: Fundus Photography — Each participant in this study will undergo fundus photography of each eye. Fundus photography involves the use of a retinal camera coupled with a low power microscope to capture photographs of the retina.
  Other Names: Photography of the Eye

SUMMARY:
Alzheimer's disease (AD) and frontotemporal dementia (FTD) are two of the most common types of age-related neurodegenerative disorders. Identifying at-risk patients and gauging disease progression in a non-invasive manner would be invaluable. Early and correct diagnosis is crucial for coordinating supportive care, patient expectations, caregiver arrangements and family planning. In addition, as treatments become available, beginning therapy early in the disease before symptoms become severe will be important. Multimodal ocular imaging (MOI) includes an ophthalmic (eye) exam and eye photographs to evaluate different layers of the retina, which is the light sensing layer of the eye. Newer technologies make it possible to visualize the disease process occurring in AD and FTD by using MOI to look at the retina, since the retina is fundamentally an outward extension of the brain itself. This study will attempt to correlate signs of disease in the retina, as determined by MOI, with plaque buildup in the brain as seen by imaging. This will demonstrate the sensitivity and specificity of MOI for diagnosing AD and FTD in a noninvasive manner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with dementia must have known diagnosis of Alzheimer's dementia (AD) or frontotemporal dementia (FTD)
* Subjects with dementia must have Moderate/severe dementia as preferentially defined by a documented MoCA score of less than 17, or by MMSE score of less than 17, within the last 12 months
* Individuals with no evidence of AD or FTD as age-matched controls.

Exclusion Criteria:

* Preexisting retinal or optic nerve disorder including macular degeneration, diabetic retinopathy, retinal dystrophy, and glaucoma
* Anterior segment abnormalities of the eye limiting ocular imaging (e.g. corneal disorders, dense cataract).
* Use of medications with known effects on the retina or optic nerve (e.g. hydroxychloroquine, ethambutol).
* Pregnant or lactating women.
* Prisoners.
* Subjects with advanced dementia who cannot be independently and reliably positioned at the ocular imaging device for reliable imaging.
* Subjects with contraindications to magnetic resonance (MR) imaging, including pacemakers or claustrophobia.
* Evidence of large vessel stroke or mass lesion identified on MR imaging.
* Subjects limited by participation in research procedures involving ionizing radiation.
* Subjects who are already participating in another clinical study or clinical trial
* Participants with a clinically significant or unstable medical or surgical condition that, in the opinion of any of the investigators, might preclude safe completion of the study or might affect the results of the study. These include conditions causing significant central nervous system or autonomic dysfunction, such as congestive heart failure, recent (<6 months) myocardial infarction, thrombocytopenia (<50 x 10(9)/L), immunosuppressed state, severe uncontrolled hypertension, severe cardiopulmonary disease, severe anemia (hemoglobin <8g/dl), severe liver or kidney disease (creatinine >2.3 mg/dl) uncontrolled diabetes mellitus (HgbA1c >10g%), alcoholism, malignant neoplasms, amyloidosis, uncontrolled hypothyroidism, unstable peripheral neuropathies, concurrent infections, orthopedic problems that compromise mobility and activities of daily living, severe cerebrovascular accidents (causing symptoms such as hemiplegia, aphasia and non-dominant parietal lobe syndrome), history of exposure to neurotoxins or neuroactive drugs, or parkinsonism due to drugs (including neuroleptics, alpha-methyldopa, reserpine, metoclopramide).

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited with mid-to-late stage AD and FTD, as well as age-matched healthy controls, using the extensive database of research participants maintained by the Michigan Alzheimer's Disease Center (MADC).
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Presence of Retinal Thinning | 45 minutes
  Imaging of the eye will be used to measure differences in retinal thickness between subjects with Alzheimer's Dementia, Frontotemporal Dementia, and healthy age-matched controls.

SECONDARY OUTCOMES:
Presence of Amyloid Plaque | 45 Minutes
  Fundus autofluorescence (FAF) will be used to detect the presence of lipofuscin
Presence of Brain Pathology | 60 Minutes
  MRI of the brain will be performed in order to determine if pathology observed on neuroimaging correlates quantitatively and/or qualitatively with retinal thickness.
Presence of Brain Metabolism | 180 Minutes
  PET scanning of the brain will be performed in order to determine if brain metabolism observed on neuroimaging correlates quantitatively and/or qualitatively with retinal thickness.
Presence of Macular Vascular Anomalies | 45 Minutes
  Imaging of the eye will be used to measure differences in vascular density between subjects with Alzheimer's Dementia, Frontotemporal Dementia, and healthy age-matched controls.

CONTACTS AND LOCATIONS:
Overall Officials: Cagri G. Besirli, MD PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD Data may be shared if requests to the PI are made, a reasonable plan is proposed, and Data Use agreements are put in place.